CLINICAL TRIAL: NCT02038803
Title: Patient Preferences and Efficacy of TOBI Podhaler vs. Tobramycin Inhalation Solution (PETIS)
Brief Title: Efficacy of TOBI Podhaler vs. Tobramycin Inhalation Solution
Acronym: PETIS
Status: Terminated | Type: Observational
Why Stopped: The project was a student driven study. The student graduated prior to the subjects completing all research related activities. As a result, the study was closed prematurely.
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Robert A Balk, Director, Division of Pulmonary and Critical Care Medicine, Rush University Medical Center
Other Study IDs: 13080201
Record Dates: First submitted 2014-01-15; First posted 2014-01-17 (Estimated); Results first posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-10

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis Medication Adherence
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adults- Cystic Fibrosis: Adults with cystic fibrosis who have respiratory colonization with Pseudomonas Aeruginosa. The actual study will involve instructing adult patients with CF on the use of a new form of Tobramycin for inhalation (powder) and then assessing this new form of TOBI podhaler vs the old TOBI solution related to patient preference on use, time involved in taking the new medication vs the old, and impact on their pulmonary function and subsequent exacerbation rate plus quality of life.
  Interventions: Drug: TOBIpodhaler

INTERVENTIONS:
Drug: TOBIpodhaler
  Other Names: Inhaled TOBI solution

SUMMARY:
Inhaled tobramycin is a Cystic Fibrosis Foundation recommended effective treatment for individuals with cystic fibrosis for the management of Pseudomonas aeruginosa airway colonization and improves the FEV1 and reduces the number of acute pulmonary exacerbations of CF. Patients typically use the inhaled tobramycin for a period of 28 days. Unfortunately, the standard nebulizer method for delivering tobramycin inhaled solution (TIS) is time-consuming and may result in missed therapy doses and suboptimal care. A new inhaled formulation and delivery device, the TOBI Podhaler (TPI), an alternative method of administering inhaled Tobramycin will be used and assessed. This new pocket-sized disposable inhaler is maintenance-free, requires no refrigeration or power source, and should greatly increase patient mobility and improve time management.

DETAILED DESCRIPTION:
Adult cystic fibrosis patients from the Rush University Medical Center Adult Cystic Fibrosis Program will be recruited for a prospective before and after cohort study to evaluate patient preference for either the TOBI Podhaler or inhaled tobramycin solution and compare the efficacy of the TOBI Podhaler to tobramycin inhaled solution. This project will evaluate the potential differences in efficacy, medication adherence, treatment time, side effects/adverse effects, quality of life, and identify patient preferences between the use of TIP and TIS. Measurements after a 28-day cycle of tobramycin inhaled solution, first 28-day cycle of TOBI Podhaler and third 28-day cycle of TOBI Podhaler will include FEV1, number of acute pulmonary exacerbations, adherence, cough frequency, sputum characteristics, and side effects or adverse events. The quality of life as assessed by the Cystic Fibrosis Questionnaire-Revised (CFQ-R) will be measured after a 28-day cycle of tobramycin inhaled solution and the third 28-day cycle of TOBI Podhaler. The FEV1 values, number of missed treatments, and total treatment time will be analyzed through a repeated measures analysis of variance. Comparisons of the CFQ-R data before and after the switch to the TPI will be made with the Student's t-test.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥ 18 years) diagnosed with cystic fibrosis
2. Airway colonization with Pseudomonas aeruginosa that is sensitive to tobramycin in vitro and currently managed with Tobramycin inhaled solution who are interested in switching to the TOBI Podhaler.

Exclusion Criteria:

1. Persons unable to communicate in English,
2. Pregnant patients,
3. Patients < 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (≥ 18 years) diagnosed with cystic fibrosis
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2013-10-10 (Actual); Primary Completion 2014-05-07 (Actual); Study Completion 2014-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Balk, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was very slow related to cost of the medication. We also experienced difficulty getting subjects to return the questionnaire related to time involved and satisfaction with the treatment.
Pre-assignment Details: Subjects were asked to compare the time and satisfaction of the TOBIpodhaler treatment to their prior inhaled antibiotic administration time and satisfaction and to compare their Quality of Life (using CFR-Q) measured before and after the TOBIpodhaler.
Period: Overall Study
Arm/Group | Adults- Cystic Fibrosis
Started | 5
Completed | 0
Not Completed | 5
Not completed — poor adherence of subjects to protocol and withdrawal from study. | 4
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: 5 individuals actually started the study and participated in the initial data collection
Groups:
- Subject Response to TOBIpodhaler Were Compared to Baseline: Individuals who were on inhaled antibiotic therapy as part of their CF management of Pseudomonas in the airway were selected if they were able to change their inhaled antibiotic to the TOBIpodhaler. These subjects would then compare their time involved in airway treatment, satisfaction with the treatment, and FEV1 to their prior-to-change value.
Arm/Group | Subject Response to TOBIpodhaler Were Compared to Baseline
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.4 (5.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Region of Enrollment [Count of Participants; unit: Participants] — U.S. adult patients using inhaled TOBI and planning to switch to TOBIpodhaler
  Participants
    United States | 5
FEV1 [Count of Participants; unit: Participants] — spirometry was performed on carefusion Vmax calibrated spirometer Population: 4 subjects did not return for evaluation
  1 subject lost to follow-up All 5 subjects did not complete the study

OUTCOME MEASURES:

1. Primary Outcome: Increased Adherence to the Medical Therapeutic Regimen
Description: Number of Participants with Adherence to Tobramycin Inhaled Solution Treatment compared with TOBI Podhaler Treatment based on improved efficacy and time required for administration and translate into improved respiratory status for adult patients with cystic fibrosis.
Time Frame: 6 months
Population: 4 of 5 patients preferred TOBIpodhaler
Measure: Number; unit: participants
Groups:
- Patient Served as Own Control: Compared time spent and FEV1 change along with survey of preference.
Arm/Group | Patient Served as Own Control
Number analyzed (Participants) | 5
participants | 4

2. Secondary Outcome: Preference for TOBIpodhaler Treatment
Description: The subject will indicate a preference for TOBIpodhaler vs prior treatment.
Time Frame: 6 months
Population: Data were not collected since patients did not return for follow-up.
Groups:
- Adults- Cystic Fibrosis: Adults with cystic fibrosis who have respiratory colonization with Pseudomonas Aeruginosa. The actual study will involve instructing adult patients with CF on the use of a new form of Tobramycin for inhalation (powder) and then assessing this new form of TOBI podhaler vs the old TOBI solution related to patient preference on use, time involved in taking the new medication vs the old, and impact on their pulmonary function and subsequent exacerbation rate plus quality of life.
  TOBIpodhaler
Arm/Group | Adults- Cystic Fibrosis
Number analyzed (Participants) | 0

3. Secondary Outcome: Spirometry Data
Description: spirometry was performed at baseline and at the end of the study.
Time Frame: 6 months
Population: Data were not collected since patients did not return for follow-up.
Arm/Group | Adults- Cystic Fibrosis
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Tobramycin Inhaled Solution: Before and after study of patients with cystic fibrosis and Pseudomonas colonization comparing the time spent with TOBIsolutions vs TOBIpodhaler. The preference was evaluated including changing lung function over the course of the study.
- TOBI Podhaler: patient with cystic fibrosis using TOBI podhaler treatment.
Arm/Group | Tobramycin Inhaled Solution | TOBI Podhaler
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

LIMITATIONS AND CAVEATS:
There was limited enrollment and lack of follow up survey completion. Study was terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No